CLINICAL TRIAL: NCT06449378
Title: Multi-center, Single-arm, Prospective Study of Transorb™ Self-Gripping REsorbable Mesh in High-risk subjeCts Undergoing Open Repair of VEntral heRnia
Brief Title: Transorb™ Self-Gripping Resorbable Mesh in High-risk Subjects Undergoing Open Repair of Ventral Hernia
Acronym: RECOVER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT21008
Record Dates: First submitted 2024-05-22; First posted 2024-06-10 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Hernia; Hernia, Ventral; Hernia, Abdominal; Hernia Abdominal Wall
Keywords: Hernia Recurrence; Hernia; Hernia, Ventral; Hernia, Abdominal; Hernia Abdominal Wall
MeSH Terms: conditions — Hernia; Hernia, Ventral; Hernia, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Hernia Repair (Experimental): single arm study, no control arm
  Interventions: Device: Transorb™ Self-Gripping Resorbable Mesh

INTERVENTIONS:
Device: Transorb™ Self-Gripping Resorbable Mesh — Self-Gripping Resorbable Mesh used for repair of open ventral hernia.

SUMMARY:
The purpose of RECOVER is to evaluate the performance and safety of Transorb™ self-gripping resorbable mesh in high-risk subjects (at least one risk factor impairing wound healing) when used for reinforcement of abdominal wall soft tissues in procedures involving open extraperitoneal ventral hernia repair, in clean (US); and clean and clean-contaminated (Europe) surgical fields (Centers for Disease Control and Prevention (CDC) Classification I and II. Data from this study will primarily be used to support market approval and European post-market clinical follow-up needs. Secondarily, data will be used for product marketing, future product development, and to support market release and maintenance in global geographies.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the performance (hernia clinical recurrence rate) of Transorb™ mesh within 12 months post-operatively when the mesh is used for repair of open ventral hernia.

The secondary objectives of the study are to evaluate the safety and performance of Transorb™ mesh when used for repair of open ventral hernia within 60 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent
2. Subject is 18 years of age or older at the time of consent
3. Subject is undergoing a planned, elective, open, single-staged repair of a midline primary or incisional ventral hernia using retrorectus/retromuscular mesh placement with or without Transversus Abdominis Release (TAR)
4. Subject is expected to meet the criteria for:

   1. In the US: a class I / clean wound as defined by the CDC (Centers for Disease Control and Prevention) wound classification
   2. In Europe: a class I / clean wound or a class II / clean-contaminated wound as defined by the CDC wound classification in compliance with these conditions:

      * No break in the sterile technique, and
      * Entry into gastrointestinal tract with no or minimal spillage
5. Subject has at least one of the following comorbid factors impairing wound healing:

   1. Current smokers (subject who has smoked 100 cigarettes in his or her lifetime and who currently smokes) Note: Use smoking status prior to preoperative optimization for inclusion assessment.
   2. Smokers with a minimum 20 pack year history (including former smokers)
   3. Obesity, defined as body Mass Index (BMI) between 30kg/m2 and 39.9kg/m2
   4. Chronic Obstructive Pulmonary Disease (COPD)
   5. Diabetes mellitus
   6. History of wound infection
   7. Malnutrition (serum albumin less than 3.4 g/d)
   8. Coronary Artery Disease (CAD)
   9. History of chemotherapy
   10. Diagnosis of hypertension
   11. History of malignancy without evidence of active disease
   12. Renal insufficiency (serum creatinine concentration ≥2.5 mg/d)

Pre-Operative Exclusion Criteria Assessed during subject screening:

1. Subject is involved in another interventional drug or device study
2. Subject is unable or unwilling to comply with the study requirements or follow-up schedule
3. Subject has a history of:

   1. Previous hernia repair involving retrorectus/retromuscular mesh placement or a component separation technique (CST)
   2. Allergic reactions to products with PLLA/TMC (Poly-L-lactide, poly-trimethylene carbonate copolymer)
   3. Solid organ transplantation
4. Subject has current diagnosis/usage of:

   1. BMI greater than or equal to 40.0 kg/m2
   2. Human Immunodeficiency Virus (HIV)
   3. Collagen formation disorder (such as Ehlers-Danlos syndrome and Marfan's syndrome)
   4. Liver cirrhosis and/or current ascites
   5. Renal disease requiring dialysis
   6. Bleeding disorder and/or cannot be removed from anticoagulants prior to surgery based on surgeon discretion and standard-of-care (excluding aspirin)
   7. Chronic immunosuppression therapy (10 mg or greater of prednisone or equivalence/ day)
   8. Current or anticipated chemotherapy/radiotherapy during study period
   9. Stoma
   10. Any systemic or local ongoing infection that is uncontrolled and/or requiring treatment such as antimicrobial medication (Note: other uses of antimicrobial medications not excluded)
5. Subject has life expectancy of less than 5 years based on the judgement of investigator
6. Subject is pregnant or is planning pregnancy within the 60-month follow-up period (females of childbearing potential will be required to provide either a urine or serum pregnancy test, except for subjects who are surgically sterile, or are at least 2 years post-menopausal)
7. Subject is breastfeeding or is planning to breastfeed during the study duration period
8. Subject has any other medical condition that precludes the subject from participation, in the opinion of the investigator
9. Subject is undergoing:

   1. Minimally invasive hernia repair (i.e., laparoscopic or robotic surgery)
   2. An emergency surgery (i.e., lifesaving procedures performed where subject is in imminent danger of death)
   3. Multi-stage hernia repair
   4. Parastomal hernia repair
   5. Concomitant ostomy (creation or closure)
   6. Any other additional anticipated surgery, if subsequent surgery that would jeopardize previous application of study device, in the opinion of the investigator

   Pre-Operative Exclusion Criteria assessed/confirmed on day of surgery:
10. Subject is American Society of Anesthesiology Class 4, 5, or 6
11. Subject has a BMI greater than or equal 40.0 kg/m2
12. Subject is pregnant or is planning pregnancy within the 60-month follow-up period (females of childbearing potential will be required to provide either a urine or serum pregnancy test, except for subjects who are surgically sterile, or are at least 2 years post-menopausal)

Intraoperative Exclusion Criteria Assessed by investigator following reduction of hernia and preparation of the retrorectus/ retromuscular space for mesh placement:

1. Subject has existing mesh from previous ventral hernia surgery that investigator was unable to completely remove
2. Subject has concomitant diastasis (>2 cm) that was not repaired
3. Hernia defect that will require a multi-stage repair
4. Subject no longer meets Inclusion Criteria 4
5. Subject who will require more than a single piece of Transorb™ or any other additional mesh
6. Subject with anticipated inability to achieve both:

   1. Midline anterior and posterior rectus fascia closure without excessive tension, and
   2. Skin closure
7. Subject who is otherwise no longer eligible to receive Transorb™ in open retrorectus/retromuscular position with or without Transversus Abdominis Release (TAR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical hernia recurrence | within 12 months
  Occurrence of clinical hernia recurrence evaluated by physical examination and confirmed, if deemed necessary by a study investigator, following site standard of care medical imaging for hernia evaluation.

SECONDARY OUTCOMES:
Rate of clinical hernia recurrence | within 1, 6, 24, 36, 48 and 60 months
  Occurrence of clinical hernia recurrence evaluated by physical examination and confirmed, if deemed necessary by a study investigator, following site standard of care medical imaging for hernia evaluation.
Rate of clinical hernia recurrence requiring re-operation | within 1, 6, 12, 24, 36, 48 and 60 months
  Occurrence of operative procedures performed with the specific goal of repairing a recurrent hernia
Time to hernia recurrence | Day 0 (day of surgery) through the 60-month visit
  Days/months to hernia recurrence measured from study procedure to clinical hernia recurrence
Rate of mesh removal related to study device and/or study procedure | within 1, 6, 12, 24, 36, 48 and 60 months
  Occurrence of study mesh removal related to study device and/or study procedure (defined as study device implantation following reduction of hernia and preparation of the retrorectus/retromuscular space)
Surgeon satisfaction | Day 0 (day of surgery)
  Surgeon satisfaction questionnaire on mesh use
Rate of surgical site occurrence (SSO) | at discharge (post-surgery up to 1-mo), and within 1, 6, 12, 24, 36, 48 and 60 months
  Occurrence of SSO defined as seroma, hematoma, wound dehiscence, or surgical site infection (SSI) that are adverse events related to study device and/or study procedure (defined as study device implantation following reduction of hernia and preparation of the retrorectus/retromuscular space)
Rate of surgical site occurrence (SSO) requiring a procedural intervention (SSOPI) | at discharge (post-surgery up to 1-mo), and within 1, 6, 12, 24, 36, 48 and 60 months
  Occurrence of SSO defined as seroma, hematoma, wound dehiscence, or surgical site infection (SSI) that are adverse events related to study device and/or study procedure (defined as study device implantation following reduction of hernia and preparation of the retrorectus/retromuscular space) and requiring a procedural intervention (defined as percutaneous drainage, wound opening or debridement, suture excision, or mesh removal (partial or total))
Hospital length of inpatient stay | discharge (post-surgery up to 1-mo)
  days spent inpatient
Rate of hernia recurrence reported by subjects | at 36, 48 and 60 months
  Occurrence of subject-reported hernia recurrence through the Ventral Hernia Recurrence Inventory (VHRI)
Change in subject quality of life (QoL) | baseline compared to 1, 6, 12, 24, 36, 48 and 60 months.
  Change in subject quality of life (QoL), as measured by the Abdominal Hernia-Q (AHQ) Quality-of-Life survey patient-reported outcome measure
Change in subject-reported pain | baseline compared to 1, 6, 12, 24, 36, 48 and 60 months.
  Change in subject-reported pain at the hernia site using a Pain Numeric Rating Scale (NRS) from 0-10, with 0 being no pain and 10 being the worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Goldblatt, MD, FACS, Study Chair — Medical College of Wisconsin; Bruce Ramshaw, MD, FACS, Study Chair; J. Scott Roth, MD, FACS, Study Chair — University of Kentucky; Frederik Berrevoet, Prof. Dr., Study Chair — University Hospital, Ghent; Yohann Renard, Prof., Study Chair — CHU de Reims
Locations (13):
- United States (6):
  - Northwestern University, Evanston, Illinois
  - University of Kentucky, Lexington, Kentucky
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - TPMG General Surgery and Hernia Center, Newport News, Virginia
- UZ Leuven, campus Gasthuisberg, Leuven, Belgium
- France (6):
  - APHP Hospital Louis Mourier, Colombes
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Centre Hospitalier Universitaire de Reims, Reims
  - Hôpital Charles Nicolle Centre Hospitalier Universitaire de Rouen, Rouen
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roth JSS, Ramshaw B, Renard Y, Passot G, Berrevoet F, Bayliss K, Blanc M, Cain C, Goldblatt M. New synthetic resorbable mesh for open ventral hernia repair: the multicentre, single-arm, prospective study of Transorb self-gripping resorbable mesh in subjects undergoing open repair of ventral hernia in clean and clean-contaminated fields (RECOVER) protocol. BMJ Open. 2025 Jul 17;15(7):e100294. doi: 10.1136/bmjopen-2025-100294. PMID 40675633